CLINICAL TRIAL: NCT04073004
Title: Rapid Resolution Therapy (RRT) for Post-traumatic Stress Disorder (PTSD) Symptoms in Survivors of Sexual Violence
Brief Title: RRT for PTSD Symptoms in Survivors of Sexual Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1453
Record Dates: First submitted 2019-08-19; First posted 2019-08-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: PTSD; Rape Sexual Assault
Keywords: PTSD; Psychotherapy; Rape
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: all participants will receive the same treatment. The investigators will compare their results to data reported by Rothbaum et al (2005) which includes 2 treatment groups and a control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rapid Resolution Therapy (Experimental): RRT is a talk therapy that uses Neurolinguistic Programming Language and trance states to cause a shift in how the mind is processing incoming data.
  The understanding is that the part of the mind that is causing the disturbing emotion, thought or sensation is causing them to cause the person to take an action to ensure the organisms survival. RRT therapists employ psycho-therapeutic techniques taht are designed to cause the mind to process information differently so that the disturbing content and distorted meaning shift.
  Interventions: Behavioral: Rapid Resolution Therapy

INTERVENTIONS:
Behavioral: Rapid Resolution Therapy — psychotherapy that includes trance states

SUMMARY:
Study to provide evidence of efficacy for Rapid Resolution Therapy in symptoms of PTSD, Anxiety, and Depression in survivors of sexual violence.

DETAILED DESCRIPTION:
The investigators will recruit 24 participants to complete pre-test measures, participate in a 3 hour therapy session of Rapid Resolution Therapy (RRT), and then re-test one week post treatment and 6 months follow up.

If participants do not report a "good result" following the 3 hour session, the investigators will offer a 1.5 hour follow up session Participants will receive free therapy for their participation, but will not be paid.

Participants will be men and women over the age of 18 who do not have a diagnosis of psychosis and are not actively suicidal and have experienced a single rape at least 3 months before enrolling in the study.

Sessions will be audio recorded and transcribed for construct validity (of RRT). Identifying in formation will be removed by the study coordinator before transcripts are coded for validity.

This study proposes to use the same methods as Rothbaum et al (2005) published in Journal of Traumatic Stress that compares Prolonged Exposure to Eye Movement and Desensitization and Reprocessing (EMDR) for PTSD Rape Victims. The investigators will compare our results to theirs. Both of their treatments were 8 sessions, and this study's treatment is one. They also include data for a control group.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* self report experiencing a rape any time before 3 months prior to treatment
* on PCL-C (Positive for PTSD)

  * score 3-5 on at least one item 1-5
  * score 3-5 on at least 3 items 6-12
  * score 3-5 on at least 2 items 13-17

Exclusion Criteria:

* history of schizophrenia or psychosis current
* suicidal risk
* in an ongoing threatening situation (i.e. domestic violence)
* participants who are pregnant or become pregnant during the study (if someone becomes pregnant during the study, we will complete treatment if she desires, but will not include data)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in The Clinician-Administered PTSD Scale (CAPS-5: Weathers et al, 2015) | pre-intervention (one month version), one week post intervention (past week version) , 6 months post intervention (one month version)
  The CAPS-5 is a 30-item structured interview that can be used to make current (past month) diagnosis of PTSD, make lifetime diagnosis of PTSD and assess PTSD symptoms over the past week In addition to assessing the 20 Diagnostic and Statistics Manual- 5th Edition (DSM-5) PTSD symptoms, questions target the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms since a previous CAPS administration, overall response validity, overall PTSD severity, and specifications for the dissociative subtype (depersonalization and derealization).
  The scale measures 1) severity of PTSD symptoms 2) severity of PTSD clusters and 3) PTSD Diagnostic status.
Change in PTSD Symptom Scale Self-Report- Civilian Version (PSS-SR: Foa et al, 1993) | screening, one week post-treatment, 6 month follow up
  A 17 item self-report measure that corresponds to the 17 DSM-IV PTSD symptoms. Items are rated 0 (not present) to 3 (very much).
  Responses create three subscales, including re-experiencing, avoidance, and arousal, as well as a total score that ranges from 0 to 51. Score above 13 indicate a presence of PTSD.
  we expect to see scores decrease post-treatment and to stay lower than baseline at 6 month follow up.
Change in Beck Depression Inventory (BDI): beck et al, 1988) | pre-intervention, one week post intervention, 6 month follow up
  The BDI is a 21 item self-report questionnaire widely used in research on depression to evaluate cognitive and vegetative symptoms of depression.
  The inventory includes 21 items rated from 0 to 3, with 0 being absence of symptoms and 3 being extreme symptoms. A score between 1 and 16 indicates a low level of mood disturbance, 17-30 indicates Moderate depression, and 31 and up indicates severe or extreme depression. We are looking for a decrease in scores with treatment, and lower than baseline score at 6 month follow up.
Change in The State Trait Anxiety Inventory (STAI: Spielberger et al, 1970) | Pre-intervention, one week follow up, 6 month follow up
  STAI is a 40-item self-report measure with two scales designed to assess state anxiety and trait anxiety.
  Items are score on a 4-point Likert scale, with 4 being most severe. 20 items measure state anxiety and 20 measure state anxiety. Scores on each scale range from 20-80, with lower scores indicating more mild anxiety and higher scores indicating clinical anxiety. We are looking for scores to go down with treatment and remain lower than baseline at 6 month follow up.

SECONDARY OUTCOMES:
Session Rating Scale (Miller et al 2002) | one week post intervention
  A 4-item continual scale measure that asks the client to report on his or her experience of the session: relationship, goals and topics, approach or method and overall from negative to positive. The rater uses a ruler to divide the scale into 10 intervals and gives the score that matches the position on a line between positive and negative
Outcome Rating Scale (ORS: Miller and Duncan, 2000) | One week post intervention
  A 4-item continual scale measure that asks the client to report on his or her subjective experience of how s/he is feeling individually, interpersonally, socially, and overall. The rater uses a ruler to divide the scale into 10 intervals and gives the score that matches the position on a line between positive and negative

CONTACTS AND LOCATIONS:
Overall Officials: Heather Aberle, MA, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado at Denver counseling center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rothbaum BO, Astin MC, Marsteller F. Prolonged Exposure versus Eye Movement Desensitization and Reprocessing (EMDR) for PTSD rape victims. J Trauma Stress. 2005 Dec;18(6):607-16. doi: 10.1002/jts.20069. PMID 16382428
- See also: cite describing RRT and link to members — http://rapidresolutiontherapy.com
- See also: site describing PCL-C and updated version — http://www.ptsd.va.gov/professional/assessment/adult-sr/ptsd-checklist.asp
- See also: Site describing CAPS-5 — http://www.ptsd.va.gov/professional/assessment/adult-int/caps.asp
- See also: Pearson Assessments site describing psychometric properties of the BDI-II — http://pearsonclinical.in/solutions/beck-depression-inventory-ii-bdi-ii/
- See also: Publisher's description and psychometric properties of the State Trait Anxiety Inventory — http://www.mindgarden.com/145-state-trait-anxiety-inventory-for-adults